CLINICAL TRIAL: NCT02603692
Title: Health Related Quality of Life in Pediatric Central Nervous System (CNS) Tumors: A Feasibility Study Utilizing PROMIS
Acronym: PROMIS-QOL
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Alex's Lemonade Stand Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: PROMIS-QOL; 2014-5742 (Other: Cincinnati Children's Hosp Med Ctr IRB#1)
Record Dates: First submitted 2015-08-03; First posted 2015-11-13 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Brain Neoplasms
Keywords: Newly diagnosed brain tumor; Progressive brain tumor; PROMIS; Quality of life
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pediatric group (ages 8-17): PROMIS pediatric domains for emotional distress (anxiety and depression), physical function (fatigue, pain interference, mobility and upper extremity), and peer relations
  Interventions: Other: PROMIS-QOL
- Adult group (ages 18-35): PROMIS adult domains. To reduce respondent burden, the multi-form design will be used which includes the short form of physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference and pain intensity.
  Interventions: Other: PROMIS-QOL
- Parent/guardian proxy: Parent/guardian will complete the parental proxy PROMIS instruments based on corresponding child age (ages 5 to 17 years)
  Interventions: Other: PROMIS-QOL

INTERVENTIONS:
Other: PROMIS-QOL — PROMIS questionnaires completed every 3 months for up to 2 years.

SUMMARY:
In this research study the investigators want to learn more about the quality of life before, during and after cancer treatment in patients with central nervous system brain tumors. Often CNS tumors and cancer treatment can cause many physical and emotional problems and side effects. Some of these problems and treatment side effects can cause a change in a patient's qualify of life and overall well-being. Quality of life questionnaires are used to measure well-being and ability to carry out daily activities by asking patients to answer several questions about their physical, emotional, and social well-being.

In this research study we want to find out if patient's answers to these questions change over the course of your treatment. We also want to see if doctors and nurses can use these answers to the questions to help patients feel better and increase their activity during cancer treatment.

DETAILED DESCRIPTION:
Pediatric CNS tumors are the second most common form of pediatric cancer and the leading cause of death related to pediatric malignancies. Over decades of work and through the efforts of collaborative groups, cure rates have increased significantly. However, various types of CNS malignancy outcomes have remained stagnant. Moreover, side effects from treatments of even the most curable CNS tumors may have dramatic short and long-term sequela ranging from cognitive, endocrine malfunction, functional mobility, neurological, and ophthalmologic compromises. As science and protocol directed therapies continue to find cures for these patients, work also must continue in efforts to explore patient reported outcomes (PROs) and health related quality of life (HRQOL) throughout the trajectory of a patient's disease process. Increased efforts in patient reported outcomes will lead to improvements in symptom management, functional status, and overall quality of life (QOL).

ELIGIBILITY:
Eligibility Criteria

* Patient must have diagnosis of a CNS tumor (newly diagnosed, relapsed, refractory, or progressed) and scheduled to receive a new therapy including surgery, chemotherapy and/or radiation therapy.
* Age: 5 -35 years of age.
* The planned therapy must include at least one disease evaluation with the first 90 days of therapy. The patient and family must intend to return to Cincinnati Children's Hospital at least once in the next 90 days.
* Each subject may only participate once in this study.
* The subject and/or his /her parent/guardian must be fluent in English. At the time of study enrollment, the medical care of the subject must be managed by an attending oncologist at Cincinnati Children's Hospital.
* The subject must have a minimum performance score of 50% (either Lansky or Karnofsky) as documented in their medical record by clinical provider (MD or nurse practitioner). Appendix I.
* A patient / family must be approached to participate in this study within 28 days of the administration of the first dose of the associated therapy or surgery.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients ages 5-35 with a diagnosis of a Central Nervous System (CNS) tumor (newly diagnosed, relapsed, refractory, or progressed) and scheduled to receive a new therapy including surgery, chemotherapy and/or radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2017-08 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of participants to complete at least 75% of the Patient Reported Outcomes Measurement Information System (PROMIS) tool in pediatric and adult patients with brain tumors. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariko DeWire, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- See also: Cincinnati Children's Cancer and Blood Diseases Institute — http://www.cincinnatichildrens.org/research/divisions/c/cbdi/default/
- See also: Cincinnati Children's Hospital Oncology Division — http://www.cincinnatichildrens.org/research/divisions/o/oncology/default/